CLINICAL TRIAL: NCT05973435
Title: Evaluation of the Level of Oxidative Stress in Relation to the Type of Anesthesia in Parturients Whose Delivery Was Completed by Caesarean Section
Status: Completed | Type: Observational
Sponsor: University Clinic Dr Dragisa Misovic-Dedinje (Other)
Responsible Party: Principal Investigator, Marina Boboš, Principal Investigator, University Clinic Dr Dragisa Misovic-Dedinje
Other Study IDs: 17/I-4
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Obstetric Anesthesia Problems
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia
  Interventions: Other: Blood sampling
- Spinal anesthesia
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sample would be taken from the participants in the study for these analyses on three occasions in 3 test tubes (before cesarean section, during cesarean section and after cesarean section).

SUMMARY:
The goal of this observational study is to assess the level of oxidative stress during cesarean section depending on the type of anesthesia applied and to determine the factors that can affect the level of oxidative stress.

The main questions it aims to answer are:

* is there any association between specific parameters of pregnancy, socio-demographic characteristics and laboratory analyses with an increased level of oxidative stress
* is there any association between type of anesthesia for ceasarean section with an increased level of oxidative stress

Blood sample would be taken from the participants in the study for these analyses on three occasions in 3 test tubes (before cesarean section, during cesarean section and after cesarean section).

Researchers will compare patients that received general anesthesia with patients under spinal regional anesthesia to see if there is any difference in level of oxidative stress measured by laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I and II

Exclusion Criteria:

* ASA status III and IV
* Emergency C section

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy pregnant women
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Elevated level of oxidative stress | 2 hours after C section
  We will measure enzymes of oxidative stress before cesarean section, during cesarean section and after cesarean section.

SECONDARY OUTCOMES:
Lactate level | 2 hours after C section
  We will measure lactate levels before cesarean section, during cesarean section and after cesarean section.
Level of cortisol | 2 hours after C section
  We will measure cortisol levels before cesarean section, during cesarean section and after cesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Center "Dr. Dragisa Misovic, Dedinje", Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No